CLINICAL TRIAL: NCT00115635
Title: A Phase I/II Study With Docetaxel and Gemcitabine in Hormonal Refractory Metastatic Prostate Cancer
Brief Title: Docetaxel and Gemcitabine in Hormonal Refractory Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Sanofi (Industry); Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UR0416; EudraCT number: 2004-002353-31
Record Dates: First submitted 2005-06-23; First posted 2005-06-24 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-10

CONDITIONS: Prostate Cancer
Keywords: Hormonal refractory, chemotherapy, docetaxel, gemcitabine
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: docetaxel
Drug: gemcitabine

SUMMARY:
The aim of the study is to determine the optimal dose of the combination of docetaxel and gemcitabine in patients with hormone refractory prostate cancer, and evaluate this dose with respect to efficacy and toxicity in a phase II trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified adenocarcinoma of the prostate.
* Hormone refractory prostate cancer (HRPC) defined as progression during previous anti-hormone treatment. Patients must have been off previous anti-androgen therapy for more than 4 weeks.
* Stage IV disease (verified by imaging or clinical examination).
* PSA > 10 microgram/l.
* PSA progression defined as a > 25% increase between two independent measurements performed with a 1-month interval or more after discontinuation of anti-androgen treatment.
* Castrate level of testosterone (< 50 ng).
* No previous oestrogen or steroid as metastatic prostate cancer treatment.
* Satisfactory hepatic function in the form of total bilirubin ≤ UNL (upper normal limit), ASAT/ALAT ≤ 2.5 x UNL, alkaline phosphatase ≤ 5 x UNL.
* Satisfactory renal function, defined as serum creatinine ≤ 1.5 x UNL.
* Satisfactory haematologic function defined as ANC >1.5 x 10^9/l, leucocytes >3.0 x 10^9/l, thrombocytes ≥ 100 x 10^9/l, haemoglobin > 7 mmol/l
* ECOG performance status ≤ 2.
* Life expectancy > 3 months.
* Patient must be able to adhere to protocol requirements.
* Written informed consent.
* > 18 years of age.

Exclusion Criteria:

* Previous prostate cancer treatment with oestrogens or steroid hormones.
* Previous chemotherapy.
* Previous treatment with systemic radioactive isotopes.
* Bisphosphonate treatment (concomitant).
* Radiation therapy covering more than 25% of the bone marrow producing area.
* Other serious coincidental and/or concomitant medical condition.
* Symptomatic cerebral metastases.
* Other previous or current malignant disease, excluding *adequately treated and cured planocellular skin carcinoma; or *other cancer assessed to carry minimal risk of recurrence.
* ECOG performance status > 2.

Ages: 18 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-03; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Prostate-specific antigen (PSA) response

SECONDARY OUTCOMES:
Clinical response
Time to PSA progression
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Sengelov, MD, Principal Investigator — Dept. of Oncology, Herlev Hospital, 2730 Herlev, Denmark
Locations (1):
- Dept. of Oncology, 54B1, Herlev Hospital, Herlev, Denmark